CLINICAL TRIAL: NCT00894010
Title: Assessment of Marketed AEDs in the Human Photosensitivity Proof of Concept Trial
Brief Title: Photosensitivity Proof of Concept Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Epilepsy Study Consortium (Other)
Collaborators: The Epilepsy Research Foundation (Unknown); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TESC-001
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Photosensitive Epilepsy
Keywords: Photosensitive epilepsy; Photosensitivity; Seizures; Epilepsy
MeSH Terms: conditions — Epilepsy, Reflex; Photosensitivity Disorders; Seizures; Epilepsy | interventions — Carbamazepine; Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: carbamazepine 400mg
  Other Names: Tegretol
Drug: levetiracetam 1000mg
  Other Names: Keppra

SUMMARY:
The purpose of this study is to determine whether patients who usually have abnormal electrical EEG responses when shown flashing lights will show a reduction in abnormal electrical activity when they take a single dose of 2 marketed drugs (carbamazepine and levetiracetam). If so, a similar study in the future may be able to identify promising new drugs for epilepsy.

Patients who successfully complete the screening visit, will return 4 additional times and will receive either placebo (2 times) or a single oral dose of both carbamazepine 400mg and levetiracetam 1000mg in random order.

During each of the study days, several procedures and intermittent photosensitivity (IPS) assessments will be performed at 5 pre-determined times over the course of the day, one pre-dose and 4 post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-60 years.
* A diagnosis and history of a photoparoxysmal response on EEG with or without a diagnosis of epilepsy for which patients are on 0-1 concomitant antiepileptic drugs.
* A reproducible IPS-induced photo-paroxysmal response (PPR) on EEG of at least 3 points on a frequency assessment scale in at least one eye condition and no change of more than 3 frequencies in 2 repeated measurements recorded at screen in at least one eye condition.
* Patients in otherwise good health (with the exception of epilepsy), as determined by the PI via the medical history, a physical examination and screening laboratory investigations.
* A body mass index (BMI) between 18 and 35.
* Able and willing to provide written informed consent to participate in the study in accordance with the ICH, GCP guidelines.

Exclusion Criteria:

* A history of non epileptic seizures (e.g. metabolic, structural or pseudo-seizures).
* Women who are pregnant or lactating.
* Women of reproductive potential who do not agree to use effective birth-control methods.
* Any clinically significant laboratory abnormality which, in the opinion of the investigator, will exclude the patient from the study.
* An active CNS infection, demyelinating disease, degenerative neurological disease or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results.
* Any clinically significant psychiatric illness, psychological or behavioral problems which, in the opinion of the investigator, would interfere with the patient's ability to participate in the study.
* Patients who have a history of seizure worsening in response to narrow spectrum drugs (including carbamazepine)
* Patients who are suffering from clinically significant active liver disease, porphyria or with a family history of severe hepatic dysfunction indicated by abnormal liver function tests greater than 3 times the upper limit of normal (AST and ALT).
* A history of alcoholism, drug abuse, or drug addiction within the past 12 months.
* Patients who have participated in any other trials involving an investigational product or device within 30 days of screening or longer as required by local regulations.
* Patients receiving more than 1 background AED for their epilepsy. Patients receiving carbamazepine for their condition.
* Patients who are allergic to levetiracetam or carbamazepine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Demonstrate the ability of carbamazepine to suppress or reduce the photosensitivity response in patients with photosensitive epilepsy. Compare the ability of carbamazepine to impact the PPR as compared with levetiracetam, which is known to suppress PPR. | At the completion of each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline French, M.D., Principal Investigator — NYU Comprehensive Epilepsy Center
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Adult Epilepsy Center, Baltimore, Maryland
  - NYU Comprehensive Epilepsy Center, New York, New York

REFERENCES:
- See also: The Epilepsy Study Consortium — http://www.epilepsyconsortium.org